CLINICAL TRIAL: NCT03350282
Title: Guanidinoacetic Acid With Creatine Compared With Creatine Alone for Tissue Bioenergetics, Hyperhomocysteinemia and Exercise Performance: a Randomized Double-blind Superiority Trial
Brief Title: Guanidinoacetic Acid With Creatine Compared With Creatine Alone for Tissue Bioenergetics, Hyperhomocysteinemia and Exercise Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSD-01
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Energy Metabolism
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mixture GAA-creatine (Experimental): Mixture of guanidinoacetic acid and creatine monohydrate
  Interventions: Dietary Supplement: GAA-creatine
- Creatine (Active Comparator): Creatine monohydrate
  Interventions: Dietary Supplement: Creatine

INTERVENTIONS:
Dietary Supplement: GAA-creatine
  Arms: Mixture GAA-creatine
Dietary Supplement: Creatine
  Arms: Creatine

SUMMARY:
Co-administration of creatine and guanidinoacetic acid (GAA) has been recently put forward as an advanced dietary strategy to optimize tissue bioenergetics. The investigators hypothesized that creatine-GAA mixture would result in more powerful rise in brain and skeletal muscle creatine, as compared to creatine supplementation alone.

DETAILED DESCRIPTION:
Targeting energy-demanding tissues in health and disease continues to be a challenging task in human nutrition and biomedicine. Impaired bioenergetics accompanies many different conditions, including cardiometabolic diseases, neurodegenerative disorders or high-intensity exercise, with various dietary interventions developed to restore cellular energy. Creatine is recognized as a beneficial and safe energy-boosting agent in both athletic and clinical environments. However, its effectiveness in specific conditions seems to be fairly restrained due to its limits in transportability and performance. Guanidinoacetic acid (GAA), a metabolic precursor of creatine, appears as a novel energy-enhancing supplement, with GAA being superior to creatine in facilitating creatine concentrations in the human brain and skeletal muscle. This perhaps happens due to GAA interaction with cellular transporters previously dismissed as untargetable carriers by other similar therapeutics. On the other hand, GAA loading remains under scrutiny due to its hyperhomocysteinemia-inducing potential, and possible neurotoxic effects. Co-administration of creatine and GAA has been recently proposed as a better strategy comparing to administration of each compound per se. Besides providing a competitive advantage for enhanced levels of tissue creatine, GAA-creatine mixture might also diminish side effects related to isolated GAA administration. However, no human studies so far evaluated the effects of this mixture. In the present study, the investigators compared the impact of 4-week co-administration of GAA and creatine vs. creatine administration alone on serum biomarkers, exercise performance and tissue bioenergetics in healthy young men.

ELIGIBILITY:
Inclusion Criteria:

* men age 18-45 years
* BMI 18.5-24.9 kg/m2
* physically active (> 150 min per week)
* free of known disease
* must be able to give written informed consent

Exclusion Criteria:

* serum homocysteine > 15 µmol/L
* use of dietary supplement (> 1 month)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Brain creatine | Baseline vs 4-week follow up
  Rise in brain creatine levels

SECONDARY OUTCOMES:
Vastus medialis creatine | Baseline vs 4-week follow up
  Rise in vastus medialis creatine creatine levels

CONTACTS AND LOCATIONS:
Overall Officials: Sergej Ostojic, MD, PhD, Study Chair — University of Novi Sad

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared via institutional repository
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available from January 2018

REFERENCES:
- [Background] Ostojic SM. Co-administration of creatine and guanidinoacetic acid for augmented tissue bioenergetics: A novel approach? Biomed Pharmacother. 2017 Jul;91:238-240. doi: 10.1016/j.biopha.2017.04.075. Epub 2017 Apr 28. PMID 28460226
- [Derived] Semeredi S, Stajer V, Ostojic J, Vranes M, Ostojic SM. Guanidinoacetic acid with creatine compared with creatine alone for tissue creatine content, hyperhomocysteinemia, and exercise performance: A randomized, double-blind superiority trial. Nutrition. 2019 Jan;57:162-166. doi: 10.1016/j.nut.2018.04.009. Epub 2018 May 17. PMID 30170305